CLINICAL TRIAL: NCT05984797
Title: Integrated Short-term Palliative Rehabilitation to Improve Quality of Life and Equitable Care Access in Incurable Cancer: A Multi-national Randomised Controlled Trial
Brief Title: Integrated Short-Term Palliative Rehabilitation in Incurable Cancer
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Hospices Civils de Lyon (Other); University of Bergen (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Research Unit for General Practice, Aarhus University (Other); University of Edinburgh (Other); EAPC (Unknown); Azienda USL - IRCCS di Reggio Emilia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INSPIRE; 328722 (Other: IRAS)
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: cancer; Rehabilitation; palliative; support; disability
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Multinational, parallel group, randomised, controlled, assessor blind, superiority trial
Who Masked: Outcomes Assessor
Masking Description: Owing to the nature of the intervention, it is not possible to blind participants or intervention practitioners. Individual participants are allocated on a 1:1 basis to receive either palliative rehabilitation plus usual care or usual care. Treatment allocation will not be disclosed to the CTRU KCTU trial team or to other members of the research teams involved in data analysis to maintain blinding during outcome assessment and to minimise possible bias. Individual participants are allocated on a 1:1 basis to receive either palliative rehabilitation plus usual care or usual care. A computer-generated minimisation programme that incorporates a random element will be used to ensure that treatment groups are well balanced for: trial country ,baseline FACT-G score (<=64, 65-79, 80+), ECOG performance status (2, 3) in order to guard against chance bias in patient allocation for prognostic factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): Integrated Short-term Palliative Rehabilitation + usual care
  Interventions: Other: Integrated Short-term Palliative Rehabilitation
- control arm (No Intervention): usual care

INTERVENTIONS:
Other: Integrated Short-term Palliative Rehabilitation — Participants will be offered up to 3 manualised sessions (face to face and/or remotely, via telephone or video-conference) delivered by an expert rehabilitation practitioner (physiotherapist, occupational therapist,).
  Core components focus on (i) self-management of symptoms, (ii) physical activities and fitness, and (iii) social participation. Delivery of rehabilitation intervention components will include explicit use of behaviour change techniques including goal setting and action planning to focus on outcomes that are meaningful for the person, their family, and clinicians.
  Arms: intervention arm

SUMMARY:
The goal of this intervention trial is to determine if palliative rehabilitation in addition to usual care is more effective than usual care at improving health-related quality of life in patients with incurable solid cancer.

DETAILED DESCRIPTION:
Background and study aims Cancer is one of the main causes of illness, burden and death in Europe. The Joint Research Centre (JRC) of the EU estimated 2.7 million new cancer cases. For all cancers, between 53-79% of men and 41-62% of women are diagnosed with incurable disease. Their cancer treatment is life-prolonging but will not cure the disease.

Cancer is also a major and growing contributor to disability (loss of function). Recent global estimates suggest a loss of 382 disability-adjusted life years per 1000 individuals. Disability is a poorly recognised and undertreated consequence of incurable cancer. Over time, loss of function results in people not being able to continue with valued roles and routines, to manage usual household and social activities, and to self-care. One-third of adults with cancer require assistance to perform basic activities like washing and dressing, and half need help with extended activities like shopping and transportation. Disability reduces quality of life and well-being. Disability related to daily activity is closely related to unplanned hospital admissions and mortality.

Palliative rehabilitation empowers people with incurable conditions to actively manage their condition themselves, enabling them to live fully and enjoy the best health-related quality of life possible, including cancer towards the end of life. It aims to reduce symptoms and help people to stay independent and socially active. WHO policy on Universal Health Coverage states both rehabilitation and palliative care as essential, quality health services. It recommends they be integrated within and between primary, secondary, and tertiary health systems using a multi-professional workforce. While integrated rehabilitation has been achieved for people with chronic respiratory, cardiac and stroke conditions, this is not the case for people with cancer, especially those living with incurable disease. Access to palliative care services has increased but access to rehabilitation remains varied.

In this study, the investigators are evaluating a rehabilitation intervention that has been designed to meet the needs of people living with advanced cancer. The study is taking place in countries across Europe, and the investigators plan to recruit 340 participants from hospitals. The investigators aim to find out if and how the rehabilitation intervention affects the participants who take part in the study. The investigators will also study how it fits in with current healthcare services.

Who can participate? This study is suitable for patients aged 18 or over, diagnosed with advanced solid cancer: lung, colorectal, breast, prostate or other, irrespective of timing in relation to any oncology or palliative care treatments.

What does the study involve? After signing the informed consent, the participation in this trial will last 16 weeks. Participation in this trial is voluntary and the participants can withdraw any time.

During the first face to face visit, participants will be randomly allocated to receive either INSPIRE rehabilitation intervention + usual care or usual care only. The random allocation will be done using a software maintained by the King's Clinical Trials Unit.

The trial schedule depends on group allocation:

Participants allocated to usual care only will be asked to complete questionnaires at weeks 4, 8 and 16 either on their own, with a help of a friend or family member, or with the researcher over the telephone or in person. It should take 30 - 45 minutes to compete all the questions.

Participants allocated to the INSPIRE rehabilitation + usual care will be offered up to 3 rehabilitation visits in addition to the questionnaire completion at weeks 4, 8 and 16. Each visit will last 30 -90 minutes.

1. st rehabilitation visit will be face to face and will be scheduled no later than 14 days after joining the trial. During this visit, a rehabilitation action plan will be put together.
2. nd rehabilitation will be scheduled around 4 weeks, but no later than 5 weeks after joining the trial.
3. rd rehabilitation visit will be scheduled around 6 weeks, but no later than 7 weeks after joining the trial.

Both visits 2 and 3 can be face to face, via telephone or via video call and participants will have the opportunity to review and, if needed, change their rehabilitation action plan.

There won't be any changes in usual care for participants that have been allocated to the rehabilitation intervention group.

Participants allocated to the INSPIRE rehabilitation intervention may also be invited to an optional one-to-one interview with a member of a research team. The interview will last around 30-60 minutes. At the week 28 the research team will look at the participants medical notes to see how they're getting on; however participants will not need to do anything at this time.

The trial team will collect participants' medical history and demographic data; however demographic data will be anonymised and only year of birth and initials will be shared with the research teams. All data will be stored on a password-protected database to which only authorised individuals will have access.

What are the possible benefits and risks of participating? The study is designed to help us understand if the rehabilitation intervention can benefit people living with advanced cancer. This is a very low risk study. This study will require attending appointments and complete questionnaires which might be tiring for some people. It is not yet clear if taking part in this study will be directly beneficial for the study participants. however, taking part should help to improve future care and research, to help care for people with similar conditions in the future.

Where is the study run from? INSPIRE is coordinated by King's College London (UK) with centres in the UK, Italy, Denmark, Norway, and France.

When is the study starting and how long is it expected to run for? September 2022 to August 2026

Who is funding the study? Funding to conduct the trial in the European Union is provided by HORIZON-HLTH-2021-DISEASE-04. In the UK this study is funded by UKRI Innovate (UKRI Reference Number: 10047799)

Who is the main contact? INSPIRE Trial Manager: INSPIRE@kcl.ac.uk

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Diagnosis of incurable solid cancer: lung, colorectal, breast, prostate or other, irrespective of timing in relation to any oncology or palliative care treatments
* Eastern Cooperative Oncology Group performance status 2-3
* Able to provide informed consent and complete trial assessments in available languages.

Exclusion Criteria:

* Blood cancers: Leukaemia, Lymphoma, Myelodysplastic Syndromes (MDS), Myeloproliferative Disorder (MPD), Multiple Myeloma.
* Currently receiving specialist rehabilitation* for their cancer or co-morbidity-related dysfunction, or received within the two weeks prior to consent.
* Clinician rated prognosis of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Assessed at 8 weeks after enrollment to the study
  Assessed using Functional Assessment of Cancer Therapy (FACT-G) General scale, where high score indicates better functional well-being and quality of life for cancer patients. Lower scores may indicate a greater burden of symptoms, reduced ability to perform daily activities, and overall lower satisfaction with life during the cancer journey.

SECONDARY OUTCOMES:
FACT-G: Assessed using Functional Assessment of Cancer Therapy - General | Assessed at 4 and 16 weeks after enrollment to the study
  Functional Assessment of Cancer Therapy (FACT) General scale at 4 and 16 weeks, where high score indicates better functional well-being and quality of life for cancer patients. Lower scores may indicate a greater burden of symptoms, reduced ability to perform daily activities, and overall lower satisfaction with life during the cancer journey.
Disability - World Health Organization Disability Assessment Schedule (WHODAS 2.0) | Assessed at 8 and 16 weeks after enrollment to the study
  Higher scores reflect more significant disability, while lower scores indicate better functional status and less disability. It is used to measure and assess the impact of health conditions or disabilities on a participant's ability to function in their daily life.
Symptoms - Palliative Outcomes Scale | Assessed at 8 and 16 weeks after enrollment to the study
  Symptoms- Palliative Outcomes Scale - Symptoms (POS-S): designed to evaluate the severity and impact of various symptoms on the participant's quality of life. Higher scores indicate more severe symptoms and a greater impact on the patient's well-being, while lower scores indicate milder symptoms and less disruption in daily life.
Goal attainment- Goal attainment scale (GAS-Light) | Assessed at 8 and 16 weeks after enrollment to the study
  Goal attainment- Goal attainment scale (GAS-Light): is a tool used to measure the extent to which an participant has achieved specific goals or objectives.
Client Service Receipt Inventory | Assessed at 8 and 16 weeks after enrollment to the study
  Client Service Receipt Inventory at 8 and 16 weeks

OTHER OUTCOMES:
Acceptability - Acceptability of Intervention Measure (AIM) and bespoke questionnaire. *Participants randomised to the intervention arm only | Assessed within first 2 weeks and then at week 8 after enrollment to the study
  Acceptability of Intervention Measure (AIM) is a 4-item scale that measures the perception of satisfaction and agreeability of an intervention. Items are rated using a Likert-type semantic differential scale, ranging from 1 to 5. The AIM has a Cronbach's alpha of 0.85
Appropriateness - Intervention Appropriateness Measure (IAM) and bespoke questionnaire. *Participants randomised to the intervention arm only | Assessed within first 2 weeks and then at week 8 after enrollment to the study
  The Intervention Appropriateness Measure (IAM), a 4-item scale measuring the perceived relevance and compatibility of the intervention. Items are rated using a Likert-type semantic differential scale, ranging from 1 to 5. The IAM has a Cronbach's alpha of 0.91
Access - semi-structured qualitative interviews | Participants will be interviewed in their own language by a researcher at the inclusion site after completing the rehabilitations intervention and their consent obtained
  Qualitative interviews will be conducted to assess the acceptability and the appropriateness of the intervention from the patients' point of view. These will allow patients to offer their opinion and feelings about the intervention, to identify convergences and divergences between the quantitative and qualitative parts, and finally to deepen our implementation evaluation of the acceptability and appropriateness aspects.
Bespoke Questionnaire. *Participants randomised to the intervention arm only | Assessed within first 2 weeks and then at week 8 after enrollment to the study
  A bespoke quantitative questionnaire was designed using adapted items from our literature review of published implementation questionnaires (https://implementationoutcomerepository.org/), rated based on a semantic differential scale (Likert-type), to fit with the ratings used for AIM and IAM

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Maddocks, Principal Investigator — KCL
Locations (11):
- Herlev Hospital, Herlev, Denmark
- Hôpital Lyon Sud HCL, Lyon, France
- Italy (2):
  - Istituto Nazionale dei Tumori di Milano, Milan
  - AUSL di Reggio Emilia, Reggio Emilia
- St Olav's Hospital, Trondheim, Norway
- United Kingdom (6):
  - Western General Hospital in Edinburgh, Edinburgh
  - St Gemma's Hospice, Leeds
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital, London
  - Worthing Hospital, Worthing
  - York and Scarborough Teaching Hospitals NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study Website — https://palliativeprojects.eu/inspire/